CLINICAL TRIAL: NCT04707625
Title: Correlation of Vascular Endothelial Growth Factor Levels in Anterior Chamber Fluid to Disease State in Patients With Retinal Vein Occlusion Receiving Standard of Care Treatment
Brief Title: Vascular Endothelial Growth Factor (VEGF) Levels in Retinal Vein Occlusion (RVO) During Anti-VEGF Treatment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: IRB stopped study due to safety concerns. No further data collection and what has been collected is not appropriate for analysis.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00064405
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2023-12

CONDITIONS: Retinal Vein Occlusion
Keywords: Vision Loss; Eye Injections
MeSH Terms: conditions — Retinal Vein Occlusion; Vision Disorders | interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: All patients will receive the same standard of care treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Aflibercept (Other): All subjects will receive aflibercept every 4 weeks. Once vascular endothelial growth factor levels become normal and macular edema improves treatment windows will be extended up to every 12 weeks.
  Interventions: Drug: Aflibercept Ophthalmic

INTERVENTIONS:
Drug: Aflibercept Ophthalmic — Anti-vascular endothelial growth factor intraocular injection
  Other Names: Eylea

SUMMARY:
The purpose of this study is to treat patients with retinal vein occlusion with standard of care anti-vascular endothelial growth factor therapy and to correlate levels of vascular endothelial growth factor in the anterior chamber fluid of the eye. This study will evaluate if measuring the vascular endothelial growth factor will help predict the timing of when anti-vascular endothelial growth factor therapy will be needed.

DETAILED DESCRIPTION:
Ten patients, 5 with branch retinal vein occlusion and 5 with central retinal vein occlusion, will receive stand of care anti-vascular endothelial growth factor over the course of 52 weeks while undergoing a paracentesis prior to each treatment. During the paracentesis anterior chamber fluid will be removed to evaluate vascular endothelial growth factor levels along with other cytokines present in the anterior chamber fluid. Ocular coherence tomography will also be collected at each visit to evaluate macular thickness which will be used to help determine treatment windows along with levels of vascular endothelial growth factor. Patients with high levels of vascular endothelial growth factor and the presence of macular edema on ocular coherence tomography will be treated every four weeks. Once vascular endothelial growth factor levels are reduced along with improvements of macula edema treatment windows will be extended to 8 weeks and then to 12 weeks once levels are normal and edema is no longer present.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to provide written informed consent.
* Diagnosis of Retinal Vein Occlusion with macular edema and central foveal thickness of greater than or equal to 300 microns confirmed by intravenous fluorescein angiography and Optical Coherence Tomography
* Visual Acuity between 20/25 and 5/200

Exclusion Criteria:

* Bilateral Retinal Vein Occlusion
* Vision worse than 5/200 in study eye
* History of myocardial infarction, ischemia, or cerebrovascular accident within 6 weeks of screening
* Concurrent Proliferative Diabetic Retinopathy and/or Maculopathy
* Concurrent Exudative Age-related Macular Degeneration
* Concurrent optic neuropathy with the presence of an afferent pupillary defect
* Previous vitrectomy in the study eye
* Currently pregnant or planning to become pregnant during the duration of the study. Women currently breastfeeding are also excluded.
* Previous treatment for retinal vein occlusion in the study eye
* Any current medical condition which, in the opinion of the investigator is considered to be uncontrolled
* History of allergy or hypersensitivity to study treatment, fluorescein, or any study procedure and treatment related ingredients (e.g. topical anesthetics, betadine, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nelson, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD at this time.

REFERENCES:
- [Background] Clark WL, Boyer DS, Heier JS, Brown DM, Haller JA, Vitti R, Kazmi H, Berliner AJ, Erickson K, Chu KW, Soo Y, Cheng Y, Campochiaro PA. Intravitreal Aflibercept for Macular Edema Following Branch Retinal Vein Occlusion: 52-Week Results of the VIBRANT Study. Ophthalmology. 2016 Feb;123(2):330-336. doi: 10.1016/j.ophtha.2015.09.035. Epub 2015 Oct 30. PMID 26522708
- [Background] Ogura Y, Roider J, Korobelnik JF, Holz FG, Simader C, Schmidt-Erfurth U, Vitti R, Berliner AJ, Hiemeyer F, Stemper B, Zeitz O, Sandbrink R; GALILEO Study Group. Intravitreal aflibercept for macular edema secondary to central retinal vein occlusion: 18-month results of the phase 3 GALILEO study. Am J Ophthalmol. 2014 Nov;158(5):1032-8. doi: 10.1016/j.ajo.2014.07.027. Epub 2014 Jul 25. PMID 25068637
- [Background] Heier JS, Clark WL, Boyer DS, Brown DM, Vitti R, Berliner AJ, Kazmi H, Ma Y, Stemper B, Zeitz O, Sandbrink R, Haller JA. Intravitreal aflibercept injection for macular edema due to central retinal vein occlusion: two-year results from the COPERNICUS study. Ophthalmology. 2014 Jul;121(7):1414-1420.e1. doi: 10.1016/j.ophtha.2014.01.027. Epub 2014 Mar 27. PMID 24679444
- [Background] Falavarjani KG, Nguyen QD. Adverse events and complications associated with intravitreal injection of anti-VEGF agents: a review of literature. Eye (Lond). 2013 Jul;27(7):787-94. doi: 10.1038/eye.2013.107. Epub 2013 May 31. PMID 23722722
- See also: Eyla prescribing information — https://www.regeneron.com/sites/default/files/EYLEA_FPI.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were inappropriately enrolled; IRB required early termination due to the number of protocol violations.
Period: Overall Study
Arm/Group | Aflibercept
Started | 17
Completed | 0
Not Completed | 17
Not completed — IRB Required Early Termination Due to Safety Concerns | 17

BASELINE CHARACTERISTICS:
Population: 10 participants appropriately consented included
Arm/Group | Aflibercept
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: IRB will not allow study team to access or analyze any data
  years | 74.4 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: IRB will not allow study team to access or analyze any data
  Participants
    Female | 6
    Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Macular Edema
Description: Measured by central retinal thickness using optical coherence tomography - OCT is an imaging method used to generate a picture of the back of the eye, called the retina. The picture is made by precisely measuring the amount of a dim red light that reflects off the retina
Time Frame: Baseline through week 35
Population: IRB terminated study early and would not allow study team to access data further.
Measure: Mean (Standard Deviation); unit: cubic microns
Arm/Group | Aflibercept
Number analyzed (Participants) | 10
cubic microns | -504.4 (300.82)

2. Primary Outcome: Change in Macular Volume
Description: as for outcome 1
Time Frame: Baseline through week 35
Population: IRB will not allow study team to access or analyze data any further.
Measure: Mean (Standard Deviation); unit: cubic microns
Arm/Group | Aflibercept
Number analyzed (Participants) | 10
cubic microns | -5.2 (4.0)

3. Primary Outcome: Change in Vascular Endothelial Growth Factor (VEGF) Level in Anterior Chamber
Description: Evaluated by Enzyme-Linked ImmunoSorbent Assay (ELISA) analysis
Time Frame: Baseline through week 35
Population: IRB will not allow study team to access or analyze data any further.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Aflibercept
Number analyzed (Participants) | 10
pg/ml | -203.5 (203.5)

4. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA)
Description: Using Snellen Visual Acuity charts - The results are based on what line the patient can read with ease - If a subject's visual acuity is so poor that the subject can't see any letters on the charts, finger counting and/or hand motions will be checked
Time Frame: Baseline through week 35
Population: IRB will not allow study team to access or analyze data any further.
Measure: Mean (Standard Deviation); unit: LOGMAR Units
Arm/Group | Aflibercept
Number analyzed (Participants) | 10
LOGMAR Units | -0.33 (0.43)

5. Secondary Outcome: Change in Intraocular Pressure (IOP)
Description: Evaluated by tonometry - Tonometry is the procedure eye care professionals perform to determine the intraocular pressure (IOP), the fluid pressure inside the eye - Most tonometers are calibrated to measure pressure in millimeters of mercury (mmHg)
Time Frame: Baseline through week 52
Population: Not measured prior to IRB-required termination
Arm/Group | Aflibercept
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Intravitreal Injections
Description: Number of injections received during study participation
Time Frame: Baseline through week 52
Population: Not measured prior to IRB-required termination
Arm/Group | Aflibercept
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Analytes - Chemokine (C-C Motif) Ligand (CCL)s
Description: Chemokine (C-C motif) ligand 2 (CCL2)/(JE/MCP-1) Monocyte chemoattractant protein 1 and C-C motif chemokine 11(CCL11)/Eotaxin - Analyzed using an ELISA multiplex
Time Frame: Baseline through week 52
Population: Not measured prior to IRB-required termination
Arm/Group | Aflibercept
Number analyzed (Participants) | 0

8. Secondary Outcome: Change in Analytes - Chemokine (C-X-C Motif) Ligand (CXCL)s
Description: CXCL1/GRO alpha/KC/Cytokine-induced neutrophil chemoattractant (CINC-1) and CXCL2/GRO beta/MIP-s/CINC-3 - Analyzed using an ELISA multiplex
Time Frame: Baseline through week 52
Population: Not measured prior to IRB-required termination
Arm/Group | Aflibercept
Number analyzed (Participants) | 0

9. Secondary Outcome: Change in Analytes - Growth Factors
Description: Epidermal growth factor (EGF) and basic fibroblast growth factor (FGF basic)/FGF2/bFGF - and Transforming growth factor alpha (TGF-alpha) - and Platelet-derived growth factor (PDGF)-AA and PDGF-AB/BBA analyzed using an ELISA multiplex Analyzed
Time Frame: Baseline through week 52
Population: Not measured prior to IRB-required termination
Arm/Group | Aflibercept
Number analyzed (Participants) | 0

10. Secondary Outcome: Change in Analytes - Interferons
Description: Interferon (IFN)-alpha 2/IFNA2, Interferon (IFN)-beta, and Interferon (IFN)-gamma - Analyzed using an ELISA multiplex
Time Frame: Baseline through week 52
Population: Not measured prior to IRB-required termination
Arm/Group | Aflibercept
Number analyzed (Participants) | 0

11. Secondary Outcome: Change in Analytes - Proteins
Description: Programmed death-ligand 1(PD-L1)/B7 homolog 1(B7-H1) Analyzed using an ELISA multiplex
Time Frame: Baseline through week 52
Population: Not measured prior to IRB-required termination
Arm/Group | Aflibercept
Number analyzed (Participants) | 0

12. Secondary Outcome: Change in Analytes - Interleukins
Description: IL-1 alpha/IL-1F1
  * IL-1 beta/IL-1F2
  * IL-1ra/IL-1F3
  * IL-2
  * IL-3
  * IL-4
  * IL-5
  * IL-6
  * IL-7
  * IL-8/CXCL8
  * IL-10
  * IL-12 p70
  * IL-13
  * IL-15
  * IL-17/IL-17A
  * IL-17E/IL-25
  * IL-33 Analyzed using an ELISA multiplex
Time Frame: Baseline through week 52
Population: Not measured prior to IRB-required termination
Arm/Group | Aflibercept
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 1 year
Description: Although the study team reported monitoring AEs during the study prior to termination, no adverse, serious adverse or mortality events were collected prior to the IRB terminating the study for safety concerns related to the conduct of the study. Termination was not due to actual adverse, serious adverse or mortality events collected.
Arm/Group | Aflibercept
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

LIMITATIONS AND CAVEATS:
IRB terminated study early due to inappropriately enrolled participants and safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT04707625/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT04707625/ICF_000.pdf